CLINICAL TRIAL: NCT07343102
Title: Incidence of Hemocompatibility Events With or Without Aspirin in Patients With CH-VAD: a Multi-centre, Observational Study
Brief Title: Incidence of Hemocompatibility Events With or Without Aspirin in Patients With CH-VAD
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Zhejiang Provincial People's Hospital (Other); Sichuan Provincial People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Shanghai Zhongshan Hospital (Other); Jiangsu Provincial People's Hospital (Other); Ruijin Hospital (Other); Sir Run Run Shaw Hospital (Other); Henan Provincial Chest Hospital (Other); Wuhan Asia Heart Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Second Hospital of Jilin University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-2961
Record Dates: First submitted 2025-11-26; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Hemocompatibility-related Adverse Event
Keywords: hemocompatibility-related adverse event

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aspirin group: Aspirin group receiving the VKA and aspirin regimen after CH-VAD implantation.
  Interventions: Device: CH-VAD
- Non-Aspirin group: Non-Aspirin group receiving the VKA without aspirin regimen after CH-VAD implantation.
  Interventions: Device: CH-VAD

INTERVENTIONS:
Device: CH-VAD — Patients who underwent CH-VAD implantation.

SUMMARY:
The goal of this observational study is to investigate the impact of oral warfarin anticoagulation combined with or without aspirin on the incidence of non-surgical hemocompatibility-related adverse events (HRAEs) and survival in advanced heart failure patients after implantation of the fully magnetic levitation left ventricular assist device (CH-VAD).

The main question it aims to answer is : The incidence of non-surgical HRAEs and survival treated with oral warfarin anticoagulation combined with or without aspirin in Chinese CH-VAD implanted advanced heart failure patients.

CH-VAD has been approved in China for the treatment of patients with advanced heart failure.

DETAILED DESCRIPTION:
This was a multi-center, retrospective observational study including patients who underwent CH-VAD implantation in 13 participating centers after its commercial approval, from Aug 2022 through Aug 2025. Patients who died during the index hospitalization were excluded. Patients whose antiplatelet regimen was modified before the occurrence of the first non-surgical hemocompatibility-related adverse event (HRAE) were also excluded to avoid exposure misclassification. Patients were divided into two groups: those receiving aspirin in addition to warfarin (ASA+VKA) versus those receiving warfarin alone (VKA only). Warfarin was started once the patient was clinically stable and able to tolerate oral medication, with a target international normalized ratio (INR) of 2.0-2.5. For patients receiving aspirin, the dose was 100 mg daily.

The primary endpoint was a composite of survival free of major nonsurgical HRAEs at 12 months. Nonsurgical events were defined as any event occurring > 14-days post implant to avoid perioperative confounding. The composite endpoint was comprised of stroke, pump thrombosis, major nonsurgical bleeding, and peripheral arterial thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent CH-VAD implantation in 13 participating centers after its commercial approval, from Aug 2022 through Aug 2025.

Exclusion Criteria:

* Patients who died during the index hospitalization.
* Patients whose antiplatelet regimen was modified before the occurrence of the first non-surgical hemocompatibility-related adverse event (HRAE) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent CH-VAD implantation in 13 participating centers during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was survival free from non-surgical HRAEs at 12 months, estimated using Kaplan-Meier methods. | Reported data includes the period from 14-days post implant to study completion. Outcome measurement is performed at the study completion, a median follow-up of 368 days.
  The composite endpoint was comprised of stroke, pump thrombosis, major nonsurgical bleeding, and peripheral arterial thromboembolism. Nonsurgical events were defined as any event occurring > 14-days post implant to avoid perioperative confounding.

SECONDARY OUTCOMES:
Secondary endpoints were the individual components of the composite. | Reported data includes the period from 14-days post implant to study completion. Outcome measurement is performed at the study completion, a median follow-up of 368 days.
  The composite was comprised of stroke, pump thrombosis, major nonsurgical bleeding, and peripheral arterial thromboembolism. Nonsurgical events were defined as any event occurring > 14-days post implant to avoid perioperative confounding.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No